CLINICAL TRIAL: NCT02293096
Title: Pharmacogenetic Prediction of Metoprolol Effectiveness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to the change in funding.
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-3174; 1K23GM110516-01 (NIH)
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
Keywords: Genotype; CYP2D6; ADRB1
MeSH Terms: conditions — Hypertension | interventions — Metoprolol; Genotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metoprolol succinate, CYP2D6 Genotyping, CYP2D6 Phenotyping (Experimental): The parent study will integrate covariates to predict metoprolol effectiveness for SBP decline of 10%. All patients will receive metoprolol. The following covariates will be used to predict metoprolol effectiveness: clinical variables (Age, sex, race/ethnicity, co-medications, and BMI) CYP2D6 genotype, CYP2D6 phenotype, and metabolomic factors.
  metoprolol succinate
  Genotyping: CYP2D6 only clinically pertinent pathway of metoprolol metabolism and polymorphisms have been associated with altered levels of metoprolol. ADRB1 is the drug target and polymorphism in this receptor has been associated with variable drug response. Genotyping will occur after the treatment phase is complete.
  CYP2D6 Phenotyping: Phenotype can be discordant from what is predicted by genotype. CYP2D6 henotyping using dextromethorphan will be used. Investigators will be blind to the patient blood pressure outcome for this intervention.
  Interventions: Drug: metoprolol succinate; Genetic: Genotyping; Procedure: CYP2D6 Phenotyping

INTERVENTIONS:
Drug: metoprolol succinate
  Other Names: Lopressor
Genetic: Genotyping — CYP2D6 only clinically pertinent pathway of metoprolol metabolism and polymorphisms have been associated with altered levels of metoprolol. ADRB1 is the drug target and polymorphism in this receptor has been associated with variable drug response. Genotyping will occur after the treatment phase is complete. Thus the investigator, the subject, and the outcomes investigator will be blind to the intervention.
  Other Names: CYP2D6 genotyping and ADRB1 genotyping
Procedure: CYP2D6 Phenotyping — Phenotype can be discordant from what is predicted by genotype due to variability in absorption, hepatic blood flow, drug interaction and drug elimination. These factors can be accounted for by utilizing a phenotyping assay that determines area under the curve of the probe since the probe is affected by the same variables dictating metabolism phenotype of the therapeutic drug. Investigators will be blind to the patient blood pressure outcome for this intervention.
  Other Names: Dextromethorphan probe of CYP2D6

SUMMARY:
The investigators will prospectively follow a population of patients with uncontrolled high blood pressure beginning metoprolol succinate therapy to determine the drug effect in an observational clinical trial. The investigators will determine each individual's genotype for both CYP2D6 and Adrenoceptor Beta 1 (ADRB1). Metabolomic markers will be identified to determine if specific metabolites are associated with drug response. The investigators' overall objective is to determine if genetics predicts metoprolol succinate response better than clinical factors such as age, race, body mass index, dose, and medication co-ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between age >30 years and < 80 years
2. Subjects have diagnosis of uncontrolled essential hypertension.

Exclusion Criteria:

1. end stage liver disease,
2. end stage renal disease,
3. pregnant females,
4. American Society of Anesthesiologists (ASA) classification of >3,
5. wards of the state, prisoners,
6. decisionally challenged,
7. HR<60 bpm,
8. AV block>240 msec,
9. active reactive airway disease,
10. illicit drug abuse in the preceding 30 days,
11. hypersensitivity to metoprolol or its derivatives
12. severe peripheral arterial circulatory disorders.

Subjects will have a screening physical exam performed by Dr. Monte prior to enrollment in the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2014-09; Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Monte, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver; Emergency Department, Aurora, Colorado, United States

REFERENCES:
- [Derived] Brocker CN, Velenosi T, Flaten HK, McWilliams G, McDaniel K, Shelton SK, Saben J, Krausz KW, Gonzalez FJ, Monte AA. Metabolomic profiling of metoprolol hypertension treatment reveals altered gut microbiota-derived urinary metabolites. Hum Genomics. 2020 Mar 11;14(1):10. doi: 10.1186/s40246-020-00260-w. PMID 32160915

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 322 participants screen failed or withdrew after consent, but prior to starting the study & receiving the intervention
Groups:
- Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping: The parent study will integrate covariates to predict metoprolol effectiveness for SBP decline of 10%. All patients will receive metoprolol. The following covariates will be used to predict metoprolol effectiveness: clinical variables (Age, sex, race/ethnicity, co-medications, and BMI) CYP2D6 genotype, CYP2D6 phenotype, and metabolomic factors.
  metoprolol succinate
  Genotyping: CYP2D6 only clinically pertinent pathway of metoprolol metabolism and polymorphisms have been associated with altered levels of metoprolol. ADRB1 is the drug target and polymorphism in this receptor has been associated with variable drug response. Genotyping will occur after the treatment phase is complete.
  CYP2D6 Phenotyping: Phenotype can be discordant from what is predicted by genotype. CYP2D6 henotyping using dextromethorphan will be used. Investigators will be blind to the patient blood pressure outcome for this intervention.
Period: Overall Study
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
Started | 140
Completed | 140
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
Number analyzed (Participants) | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.12 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 116
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 60
  White | 70
  More than one race | 6
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 140

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Decline
Description: Participants with at least a 10% decrease in SBP
Time Frame: 4-6 weeks status post initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
Number analyzed (Participants) | 140
Participants | 85

2. Secondary Outcome: Heart Rate Decline
Description: 10 % decline from pre-initiation heart rate will considered a HR decline success. Number of of participants with at least 10% decline is reported.
Time Frame: 4-6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
Number analyzed (Participants) | 140
Participants | 67

3. Secondary Outcome: Adverse Drug Events: CYP2D6 Metabolizer Status
Description: Occurrence of adverse drug events will be captured and stratified by CYP2D6 metabolizer status (Poor Metabolizer (PM), Extensive Metabolizer (EM), Intermediate Metabolizer (IM), and Ultra rapid Metabolizer).
Time Frame: 6 weeks
Measure: Number; unit: participants with events
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
Number analyzed (Participants) | 140
participants with events
  CYP2D6 metabolizer status: EM | 3
  Other Metabolizer Statuses | 0

4. Other Pre Specified Outcome: Metabolomic Factors
Description: The top 5 metabolomic factors associated with SBP decline will be captured and stratified by CYP2D6 genotype and phenotype groups.
Time Frame: 0-6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Adverse Drug Events: ADRB1 Genotype
Description: Occurrence of adverse drug events will be captured and stratified by ADRB1 genotype (strong responder, good responder, non-responder).
Time Frame: 6 weeks
Measure: Number; unit: participants with events
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
Number analyzed (Participants) | 140
participants with events
  ADRB1 genotype: Strong Responder | 1
  ADRB1 genotype: Good Responder | 2
  ADRB1 genotype: Non-responder | 0

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | Metoprolol Succinate, Genotyping, Clinical Factors, and Phenotyping
All-Cause Mortality (participants affected / at risk) | 0/140
Serious Adverse Events (participants affected / at risk) | 0/140
Other Adverse Events (participants affected / at risk) | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02293096/Prot_SAP_000.pdf